CLINICAL TRIAL: NCT05519007
Title: Clinical Evaluation of the Rate of Total Joint Infection 90-day After Surgery Following Irrigation With Next Science No-Rinse Solution vs SOC Alone
Brief Title: Rate of Total Joint Infection 90-day After Surgery Following Irrigation With Next Science No-Rinse Solution vs SOC Alone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Next Science TM (Industry)
Responsible Party: Principal Investigator, Giles Scuderi, Orthopaedic Surgery, Joint Reconstruction, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-1026
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Joint Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Next Science treatment (Experimental): The surgical site will be irrigated with NS prior to closure, which will be suctioned at the end of the treatment time
  Interventions: Other: No-Rinse Solution (NS)
- Standard of Care (Active Comparator): Saline irrigation
  Interventions: Other: Saline irrigation

INTERVENTIONS:
Other: No-Rinse Solution (NS) — The surgical site will be irrigated with NS prior to closure,
  Arms: The Next Science treatment
Other: Saline irrigation — The surgical site will be irrigated with Saline
  Arms: Standard of Care

SUMMARY:
A prospective, single-site, double-arm, parallel, interventional, randomized, controlled clinical trial to assess 90-day rate of joint infections in subjects undergoing primary hip replacements after administration of Next Science No-Rinse Solution (hereby referred to as NS) vs SOC (saline irrigation). The Next Science treatment arm will exhibit greater reduction in rate of 90-day post-operative joint infection than SOC (saline) arm

ELIGIBILITY:
Inclusion Criteria:

1. Adult that meets at least one of the below criteria at time of screening:

   * American Society of Anesthesiologists (ASA) 3 2
   * BMI >35
   * Patient with functional limitations as a result of disease1:

     * Poorly treated hypertension
     * Poorly treated diabetes
     * Chronic renal failure
     * Bronchospastic disease
     * Disease with intermittent exacerbations
     * Stable angina
     * Implanted pacemaker
   * Known history as an active nicotine use (smoker)
   * Known history of uncontrolled diabetes mellitus (HgbA1C > 7.0)
   * Known history of end stage organ disease
   * Known history of inflammatory arthritis and currently on rheumatological medication (DMARDs)
   * Known history of current active cancer treatment (chemotherapy)
   * Venous Disease (Surgical Risk Calculator from ACS-NSQIP)
   * Charleston Comorbidity Score > 2
   * Elixhauser Score >11
   * Age 65 or older
2. Subject is scheduled to primary joint replacement.
3. Subject is willing and able to comply with all study procedures including transportation to the study site for all scheduled visits and be available for the duration of the study.
4. Subject has understood, signed, and dated the informed consent form.

Exclusion Criteria:

1. Unable to provide signed and dated informed consent.
2. Unable or unwilling to comply with all study-related procedures.
3. Known history of allergic reaction to any of the study products or its components, including any products used for standard of care (such as dressings or any coverings)
4. Subject has contraindications to general anesthesia
5. Any subject positive for Covid-19 virus at time of surgical screening
6. Subjects have evidence of prolonged QT segment, per EKG.
7. Subjects from a vulnerable population, in accordance with 45 CFR 46 Subparts B, C, and D

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 936 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
infection rate | at 90 days
  Joint infection rate after surgery

SECONDARY OUTCOMES:
QT prolongation | up to 24 hours (from the time of irrigation to closure)
  Incidences of QT prolongation and short-term hypocalcemia

CONTACTS AND LOCATIONS:
Overall Officials: Giles Scuderi, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Lenox Hill Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gronbeck C, Cote MP, Lieberman JR, Halawi MJ. Risk stratification in primary total joint arthroplasty: the current state of knowledge. Arthroplast Today. 2019 Feb 5;5(1):126-131. doi: 10.1016/j.artd.2018.10.002. eCollection 2019 Mar. PMID 31020036
- [Background] Doyle DJ, Goyal A, Bansal P, et al. American Society of Anesthesiologists Classification. [Updated 2020 Jul 4]. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2020 Jan-. Available from: https://www.ncbi.nlm.nih.gov/books/NBK441940/
- [Background] Moonesinghe SR, Mythen MG, Das P, Rowan KM, Grocott MP. Risk stratification tools for predicting morbidity and mortality in adult patients undergoing major surgery: qualitative systematic review. Anesthesiology. 2013 Oct;119(4):959-81. doi: 10.1097/ALN.0b013e3182a4e94d. PMID 24195875
- [Background] Bilimoria KY, Liu Y, Paruch JL, Zhou L, Kmiecik TE, Ko CY, Cohen ME. Development and evaluation of the universal ACS NSQIP surgical risk calculator: a decision aid and informed consent tool for patients and surgeons. J Am Coll Surg. 2013 Nov;217(5):833-42.e1-3. doi: 10.1016/j.jamcollsurg.2013.07.385. Epub 2013 Sep 18. PMID 24055383